CLINICAL TRIAL: NCT04059991
Title: Antibodies in Repeated Influenza Vaccination (ARIVA) Study
Acronym: ARIVA
Status: Completed | Type: Observational
Sponsor: University Hospital, Basel, Switzerland (Other)
Collaborators: University of Oslo (Other); University of Oxford (Other); Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA) (Other)
Responsible Party: Principal Investigator, Christoph Berger, Principal Investigator, University Hospital, Basel, Switzerland
Other Study IDs: ARIVA_me17Berger
Record Dates: First submitted 2019-08-15; First posted 2019-08-16 (Actual); Last update posted 2021-09-28 (Actual); Status verified 2020-11

CONDITIONS: Vaccine Response Impaired
MeSH Terms: interventions — Influenza Vaccines

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Peripheral blood mononuclear cells, serum and RNA is collected
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Biological: Influenza Vaccination — Only subjects vaccinated against influenza will be enrolled. The study itself is observational

SUMMARY:
Viruses with high mutation rates, such influenza or HIV, pose a major challenge for vaccine design. The current influenza vaccination strategy of yearly vaccination with adapted strains aims to maximally diversify the antibody immune response to prevent viral escape. There is, however, growing evidence, that repeated vaccination with very similar viral proteins might limit, instead of broaden, diversification and thereby reduce vaccine efficacy.

The ARIVA Study prospectively studies the immunological impact of repeated influenza vaccination on viral variant recognition and antibody responses in healthy subjects cross-sectionally and over three consecutive vaccination seasons.

ELIGIBILITY:
Inclusion Criteria:

* influenza vaccination (QIIV) independent of the study
* age >18 yo

Exclusion Criteria:

* no vaccination
* current acute illness

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Healthy volunteers
Sampling Method: Non-Probability Sample
Enrollment: 150 (Actual)
Dates: Start 2017-11-01 (Actual); Primary Completion 2021-03-31 (Actual); Study Completion 2021-03-31 (Actual)

PRIMARY OUTCOMES:
Influenza specific Antibody Responses | Change between baseline and 28 days post-vaccination will be compared
  Hemagglutination titers against different H3N2 Influenza strains will be measured and compared between study subjects stratified by number of previous vaccinations

SECONDARY OUTCOMES:
Plasmablast generation | Day 7 post-vaccination
  Frequency of plasmablasts in the peripheral blood will be assessed and compared between study subjects stratified by number of previous vaccinations
BCR Repertoire composition | Cross sectional comparison of the BCR repertoire characteristics day 0 and day 28
  Sorted B cell subsets will be sequenced to define the BCR repertoire. Subjects will be compared stratified by vaccination status

CONTACTS AND LOCATIONS:
Overall Officials: Christoph T Berger, MD, Principal Investigator — University Hospital Basel, Medical Outpatient Clinic
Locations (1):
- University Hospital Basel, Basel, Switzerland

IPD SHARING:
Plan to Share IPD: Undecided